CLINICAL TRIAL: NCT06395480
Title: Albumin Utilization for Intravascular Volume Replacement in Adult Cardiac Surgical Patients : A Multicentre Prospective Cohort Study
Brief Title: Albumin Utilization in Adult Cardiac Surgical Patients : A Multicentre Prospective Cohort Study
Acronym: AlbACS-1Pro
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Kingston Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5261
Record Dates: First submitted 2024-02-21; First posted 2024-05-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Antithrombin III Levels; Albumin Levels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: All consenting adults undergoing cardiac surgery at Toronto General Hospital and Kingston Health Sciences Centre.

SUMMARY:
The goal of our proposed multicentre prospective cohort study is to characterize perioperative usage patterns of crystalloids and albumin, as well as key patient outcomes, in cardiac surgical patients. Results obtained from this observational study will be combined with the results of other studies to clarify the optimal role of albumin and other blood products in the perioperative management of cardiac surgical patients. This study will also address numerous other knowledge gaps in the area of perioperative blood product management and fluid administration in cardiac surgery and define a collaborative group to support future research in this field.

DETAILED DESCRIPTION:
This is a prospective observational study of 100 patients undergoing cardiac surgery, with a target of 50 participants per site. There is a clear need for a large-scale, multicentre, randomized trial to determine the role of albumin in cardiac surgical patients, particularly in higher risk cohorts such as patients with poor ventricular function and those undergoing complex procedures. A major obstacle to conducting this trial is a lack of data regarding perioperative albumin prescribing across providers and centres, including the indication for use, timing, formulation, and dose used in different settings (i.e., in the operating room, in the intensive care unit, and on the ward). Additionally, there is little data describing variability in typical resuscitation practices, and whether centre-level differences are associated with patient outcomes. This information is critical to inform trial design, including clinically relevant trial arms and endpoints. Thus, the goal of the proposed research is to obtain information on albumin use in cardiac surgical patients across Canada that will contribute to the design of a definitive randomized controlled trial in this population.

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥18 years old) patients undergoing cardiac surgery (with or without the use of cardiopulmonary bypass) will be eligible.

Exclusion Criteria:

* Patients who are unable to consent to the study or who refuse participation will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 100 adult (≥18 years old) patients who are undergoing major cardiac surgery. All adult (≥18 years old) patients who are undergone cardiac surgery (with or without the use of cardio-pulmonary bypass) will be eligible. There are no specific exclusion criteria, except lack of consent.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Albumin (g/L) | On CPB, in the operating room but not during CPB, in the ICU, on the ward to post operative day 28
  Type, dose and timing of administration, the setting in which it was ordered, indication for use, and the type of provider responsible for the patient at administration (surgeon, anesthesiologist, intensivist, nurse practitioner).
Antithrombin III (g/L) | On CPB, in the operating room but not during CPB, in the ICU, on the ward to post operative day 28
  Measured in g/L
Crystalloid | On CPB, in the operating room but not during CPB, in the ICU, on the ward to post operative day 28.
  and others), as well as the setting of administration will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, MD MSc FRCPC, Principal Investigator — Toronto General Hospital - University Health Network
Locations (2):
- Canada (2):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Toronto General Hospital - University Health Network, Toronto, Ontario